CLINICAL TRIAL: NCT05342181
Title: Comparison of Static and Dynamic Core Stability Exercises on Pain and Disability in Postpartum Back Pain
Brief Title: Static and Dynamic Core Stability Exercises in Potpartum Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RiphahIU Saba Amjad
Record Dates: First submitted 2022-02-20; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Back Pain
Keywords: Pain and disability in postpartum
MeSH Terms: conditions — Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static exercises (Experimental): static exercises i.e traditional exercises along with base line treatment of TENS and hot pack
  Interventions: Other: Static exercises
- Dynamic exercises (Experimental): dynamic (Swiss ball) exercises along with base line treatment of TENS and hot pack
  Interventions: Other: Dynamic exercises

INTERVENTIONS:
Other: Static exercises — Participants will be treated with static core muscle exercises that are traditional group of exercises :
  1. supine bridge
  2. plank
  3. oblique crunch
  4. side lying with Abduction
  This program includes static exercises performed thrice a week for 4 weeks.This exercise comprises 5 minutes warm up and slight stretching.Rest time of 2-3 minutes with proper stretching in between sets of activity. Subjects will be requested to undertake cool down exercises, which include aerobic workouts followed by stretching exercises, at the end of each day's exercise programme. Before beginning the next session's training, the subjects will be asked if they had any discomfort.
  Arms: Static exercises
Other: Dynamic exercises — Participants will be treated with dynamic core muscle exercises that were swiss ball exercises
  1. bridging
  2. straight leg raise in prone lying
  3. straight leg raise with hand raise in prone lying
  4. pelvic tilts
  This program includes static exercises performed thrice a week for 4 weeks.This exercise comprises 5 minutes warm up and slight stretching.Rest time of 2-3 minutes with proper stretching in between sets of activity. Subjects will be requested to undertake cool down exercises, which include aerobic workouts followed by stretching exercises, at the end of each day's exercise programme. Before beginning the next session's training, the subjects will be asked if they had any discomfort.
  Arms: Dynamic exercises

SUMMARY:
To compare the effects of static exercises with dynamic core stability on pain and disability in postpartum back pain.

DETAILED DESCRIPTION:
The study comprised 28 participants. The individuals were subdivided into binary groups, group A performed static exercises and group B performed dynamic exercises including swiss ball, each containing 14 subjects. Baseline treatment (Hot pack, TENS and posture correction) to both groups was given along with core stability exercises. Core stability exercises were performed on both group for 4 weeks. The pretreatment and post treatment tests are measured using the scale VAS (visual analog scale) and Oswestry disability index questionnaire. Both groups have shown the improvement in postpartum lumber pain and an improved in daily life activities. But swiss ball exercises have more significant improvement on pain and disability in patients having postpartum lumber pain.

ELIGIBILITY:
Inclusion Criteria:

* Age groups of 18 to 35
* Pain more than 4/10 on VAS
* Without referred pain to lower limbs
* Women with normal delivery

Exclusion Criteria:

* Nulliparous women
* Osteoporosis and OA
* Systemic arterial hypertension
* Hypersensitivity to electrical modalities
* Any fracture (spine, rib) or injury
* Any abdominal surgery
* Any other general ailment
* Vertebral or disc pathologies

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Age groups of 18 to 35 Without referred pain to lower limbs Women with normal delivery
Enrollment: 31 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | 4th week
  Oswestry disability index (ODI) is used to measure disability. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
visual analog scale | 4th week
  Visual analog scale (VAS) is usd to measure pain intensity. The findings suggested that 100-mm VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Aabroo, pp-dpt, Principal Investigator — General hospital lahore
Locations (1):
- General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No